CLINICAL TRIAL: NCT06738251
Title: A Randomized, Open-label, Controlled, Multicenter Phase III Clinical Study of SHR-A2102 for Injection Versus Investigator-selected Therapy in Locally Advanced or Metastatic Urothelial Carcinoma Previously Treated With Platinum-Containing Chemotherapy and PD-(L)1 Inhibitors and With or Without ADC
Brief Title: A Phase III Study of SHR-A2102 Versus Investigator-selected Therapy in Advanced Urothelial Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-301
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-03

CONDITIONS: Advanced Urothelial Carcinoma
MeSH Terms: interventions — Injections; Docetaxel; Paclitaxel; Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A2102 group (Experimental)
  Interventions: Drug: SHR-A2102 for Injection
- Investigator-selected therapy group (Active Comparator)
  Interventions: Drug: Docetaxel Injection; Drug: Paclitaxel Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Pemetrexed Disodium for Injection

INTERVENTIONS:
Drug: SHR-A2102 for Injection — SHR-A2102 for Injection.
  Arms: SHR-A2102 group
Drug: Docetaxel Injection — Docetaxel Injection.
  Arms: Investigator-selected therapy group
Drug: Paclitaxel Injection — Paclitaxel Injection.
  Arms: Investigator-selected therapy group
Drug: Gemcitabine Hydrochloride for Injection — Gemcitabine Hydrochloride for Injection.
  Arms: Investigator-selected therapy group
Drug: Pemetrexed Disodium for Injection — Pemetrexed Disodium for Injection.
  Arms: Investigator-selected therapy group

SUMMARY:
To evaluate the efficacy and safety of SHR-A2102 for injection versus Investigator-selected Therapy in patients with Locally advanced or Metastatic Urothelial Carcinoma who have been previously treated with platinum-based chemotherapy and PD-(L)1 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this clinical study, understand the study procedures and be able to sign the informed consent form in writing.
2. 18 to 80 years old (including boundary value), gender is not limited.
3. ECOG performance status score of 0 or 1.
4. Estimated survival ≥ 3 months.
5. Pathologically confirmed urothelial carcinoma confirmed by imaging or other methods as locally advanced unresectable or metastatic disease.
6. Patients with locally advanced or metastatic disease who have previously received both a platinum-based chemotherapy regimen and a PD-(L)1 inhibitor; patients who received platinum-based chemotherapy and/or a PD-(L)1 inhibitor as neoadjuvant or adjuvant therapy and experienced recurrence or progression during treatment or within 6 months after completing treatment will be considered to have received these therapies in the locally advanced/metastatic setting.
7. Imaging-confirmed disease progression during or after treatment with the most recent regimen.
8. Able to provide preserved or fresh tumor tissue.
9. Must be present with at least one measurable lesion according to RECIST v1.1 criteria.
10. Good level of organ function.
11. Male subjects whose partners are women of childbearing potential and female subjects of childbearing potential must use highly effective contraception from the time of signing the informed consent form until 8 months after the last dose of the trial drug.

Exclusion Criteria:

1. Planned to receive any other anti-tumor therapy during this trial.
2. Receipt of other unmarketed clinical trial drugs or treatments within 4 weeks prior to randomization.
3. Received systemic anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, targeted therapy, or immunotherapy within 4 weeks prior to randomization, and palliative radiotherapy or local therapy within 2 weeks prior to the first use of the investigational drug.
4. Prior receipt of antibody-drug conjugates containing topoisomerase I inhibitors in the composition.
5. For locally advanced or metastatic disease: patients who have previously received more than three lines of systemic therapy in this setting.For neoadjuvant or adjuvant therapy: if the disease recurs or progresses during treatment or within 6 months after its completion, the patient is considered to have received first-line systemic therapy for locally advanced or metastatic disease.
6. Prior treatment with more than 1 antibody-drug conjugate.
7. Major surgery other than diagnosis or biopsy within 4 weeks prior to randomization that requires elective surgery during the trial.
8. Received systemic glucocorticoids (prednisone > 10 mg/day or equivalent dose) or other immunosuppressants within 14 days prior to the first use of investigational drug or randomization for immunosuppressive purposes.
9. Adverse events from prior antineoplastic therapy did not recover to Grade ≤1 according to NCI-CTCAE v5.0.
10. Inadequately treated central nervous system (CNS) metastases, or the presence of uncontrolled or symptomatic active central nervous system metastases. CNS metastases that have been adequately treated and whose neurological symptoms are able to return to baseline at least 4 weeks prior to randomization (with the exception of residual signs or symptoms associated with CNS treatment) may be enrolled in the study.
11. Subject has a serous effusion with clinical symptoms or requiring puncture and drainage.
12. Any malignancy diagnosed within 5 years prior to randomization (calculated from the date of the last anti-tumor treatment), except:Localized, low-risk prostate cancer.Papillary thyroid carcinoma, basal-cell carcinoma, or squamous-cell carcinoma of the skin that has been adequately treated and shows no evidence of disease.Other carcinomas in situ that have been adequately treated and show no evidence of disease recurrence.
13. History of interstitial pneumonitis/interstitial lung disease or non-infectious pneumonitis (e.g., radiation pneumonitis) that required systemic corticosteroid therapy.Current evidence, in the investigator's judgment, of uncontrolled interstitial pneumonitis/interstitial lung disease, non-infectious pneumonitis, or any other active pneumonitis.
14. Severe infections requiring intravenous antibiotics, antivirals, or antifungals for control.
15. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
16. Has a history of immunodeficiency or organ transplantation.
17. Any serious arterial or venous thrombotic event within 6 months before randomization.
18. Those who have had significant clinically significant bleeding symptoms within 3 months before the first study drug.
19. Glycosylated hemoglobin (HbA1c) ≥8%.
20. Have severe cardiovascular and cerebrovascular diseases.
21. Allergic reaction to any component of this study treatment.
22. Female subjects who are pregnant or plan to become pregnant during the study.
23. According to the judgment of the investigator, there are concomitant diseases (such as thyroid disease and mental illness, etc.) or any other conditions that seriously endanger the safety of the patient, or affect the patient's completion of this study.
24. Prior treatment for urothelial carcinoma with all chemotherapy agents included in the control-arm regimen.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 1.5 years.
Overall Survival (OS) | Up to approximately 1.5 years and 2 years.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 1.5 years and 2 years.
Disease Control Rate (DCR) | Up to approximately 1.5 years and 2 years.
Duration of Response (DoR) | Up to approximately 1.5 years and 2 years.
Serum concentrations of SHR-A2102 | Up to approximately 2 years.
Serum concentrations of SHR-A2102 toxin | Up to approximately 2 years.
Anti-SHR-A2102 antibody (ADA) | Up to approximately 2 years.
Anti-SHR-A2102 neutralizing antibody (NAb) | Up to approximately 2 years.
Incidence and severity of adverse event (AE) | Up to approximately 2 years.
Incidence and severity of serious adverse event (SAE) | Up to approximately 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided